CLINICAL TRIAL: NCT05163106
Title: Presurgical Treatment With Ribociclib and Letrozole in Patients With Locally Advanced Breast Cancer: the NEOLETRIB Study.
Brief Title: Neoadjuvant Treatment of Locally-advanced Breast Cancer Patients With Ribociclib and Letrozole
Acronym: NEOLETRIB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: Novartis (Industry); Vestre Viken Hospital Trust (Other)
Responsible Party: Principal Investigator, Jurgen Geisler, Chief Physician, University Hospital, Akershus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021/193780(REK)
Record Dates: First submitted 2021-08-13; First posted 2021-12-20 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer; HER2-negative Breast Cancer; ER-positive Breast Cancer; Locally Advanced Breast Cancer; Luminal A Breast Cancer; Luminal B Breast Cancer
Keywords: Breast Cancer; Letrozole; Ribociclib; Combination Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Tablets; ribociclib; Goserelin

STUDY DESIGN:
Intervention Model Description: Multicentre, single-arm, open-label, neoadjuvant study model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ribociclib and Letrozole Arm (Experimental): Patients entered into this study will be given letrozole (FemarTM) in combination with ribociclib (KisqaliTM) for at least 6 months. Premenopausal women will also receive treatment with goserelin 3.6 mg s.c. every 4 weeks.
  Interventions: Drug: Letrozole 2.5mg oral tablet; Ribociclib 600mg oral tablet; Drug: Goserelin

INTERVENTIONS:
Drug: Letrozole 2.5mg oral tablet; Ribociclib 600mg oral tablet — Patients will be given letrozole 2.5mg and ribociclib 600mg daily, per oral for a period of 21 days followed by 7 days of letrozole only.
  Other Names: Femara; Kisqali
Drug: Goserelin — Premenopausal women will be given goserelin 3.6 mg (subcutaneous) every 4 weeks in concert with their Letrozole and Ribociclib treatment.
  Other Names: Zoladex

SUMMARY:
Patients with locally advanced (stage III) breast cancer (LABC) are characterized by a significantly worse prognosis compared to patients with primarily operable breast cancer. While neoadjuvant chemotherapy has been the first choice in this situation for several decades, recent evidence suggests that some patients may experience an extraordinary effect from neoadjuvant endocrine treatments involving aromatase inhibitors as monotherapy or in modern drug combinations.Selected LABC patients admitted for treatment will be offered combination therapy including letrozole and ribociclib. The overall goal of the project is to improve understanding of tumor responses and resistance in patients suffering from ER-positive/HER-2 negative locally advanced breast cancer, focusing on the role of the immune system including the gut microbiome.

DETAILED DESCRIPTION:
Neoadjuvant endocrine therapy (NET) offers a good treatment option to reduce the size of large (inoperable) primary breast tumors and/or advanced axillary lymph node metastasis prior to definite surgery. For selected patients (postmenopausal women with ER-positive breast cancer), primary endocrine therapy has been shown to be as effective as standard neoadjuvant chemotherapy. It is the general opinion that aromatase inhibitors of the "third-generation" (letrozole, anastrozole, exemestane) are the preferable drugs for neoadjuvant endocrine therapy in ER-positive, postmenopausal breast cancer patients. Anastrozole, letrozole and exemestane have been shown to suppress total body aromatisation as well as plasma and tissue estrogen levels by > 90% in vivo. All three drugs are currently used as standard care in the neoadjuvant, adjuvant and metastatic setting worldwide, including in Norway.

In 2015, a new class of anti-cancer drugs was introduced known as cyclin-dependent kinase 4 and 6 (CDK4/6) inhibitors. Following pivotal trials showing dramatic effects when combined with aromatase inhibitors or steroidal antiestrogens like fulvestrant, these compounds are now well established in distinct combinations during therapy for metastatic breast cancer. All in all, the addition of a CDK4/6 inhibitor to standard anti-hormone therapy for breast cancer doubled the time to disease progression and caused significant improvements in overall survival. Based on these findings, CDK4/6 inhibitors have also been tested in the neoadjuvant setting in clinical trials with very promising results. However, the combination of an aromatase inhibitor and a CDK4/6-inhibitor is not currently approved as standard neoadjuvant treatment for patients with locally advanced breast cancer (LABC) in Norway. Thus, the study described here will make this highly promising drug combination available for all patients who participate in this study. At the same time, the protocol will allow investigators to optimize the selection of patients benefitting from this treatment, highlight relevant biomarkers for personalized medicine and treatment, evaluate predictive markers and study the basic biology underlying treatment effects and resistance.

In recent years researchers have noted a growing body of evidence concerning the involvement of the immune system in the onset and prognosis of breast cancer both locally (in the tumor or connected tissues) and through the involvement of the immune system as a whole. Interestingly, the gastrointestinal (gut) microbiota seems to play an important role in determining whether the immune system is able to fight against several cancer types. Pre-clinical studies have shown that the microbes in the gut may influence the repertoire and activity of immune cells, such as T cells, potentially priming the immune system for cancer cell recognition and destruction. This hypothesis is supported by the finding that treatment responses to immune checkpoint inhibitors (ICIs) in a variety of cancer types is dependent on the distinct gut microbiome of an individual patient as the efficacy of the ICIs relies on the presence of cancer-recognizing T cells.

In addition, recent findings indicate that an emerging group of small molecules / targeting cancer therapies have immune altering properties. The MAPK kinase (MEK) inhibitors exemplify this by contributing to anti-tumor immunity through increasing the levels of cytotoxic T lymphocytes in preclinical model systems. Similar findings have recently been reported for both CDK4/6 inhibitors and PI3K-inhibitors. Thus, CDK4/6 inhibitors are believed to increase the antigen presentation of cancer cells, increase the activity of tumor infiltration by CD45+ cells and effector T cell activation, as well as decreasing Treg cell proliferation. While these mechanisms have been well described in in vitro and animal models, they need to be studied in humans as soon as possible to understand them and allow investigators to take advantage of these novel aspects in clinical decision making. These findings may also pave the way for microbiome and immune-related data to be used as potential biomarkers for patient selection and response evaluations during therapy.

In addition to the clinical effects of being the standard care for breast cancer patients suffering from locally advanced breast cancer, neoadjuvant therapy is widely used to study the endocrinology of breast cancer in general and is recognized as one of the best model systems to predict responses in other clinical settings (early breast cancer or metastatic breast cancer). Tumor biopsies obtained before initiation of treatment and following six months of therapy will allow correlations to the individual type of clinical response (partial responses vs complete responses etc.). The research will focus on intratumoral mechanisms of adaption through tumor characterization using single cell technology which will allow investigators to follow both the different cancer clones as well as the evolution of different immune cells during therapy. Investigators will use novel approaches to evaluate liquid biopsies (measurement of cytokines levels, metabolites and cell free DNA-fragments etc.) during letrozole and ribociclib therapy using state of the art laboratory methods available at the host hospital and in the laboratories of the listed collaborators.

Thus, all in all, the planned study will be able to contribute to the basic understanding of this very potent new drug combination that may be used in large groups of breast cancer patients in the future, including locally advanced breast cancer, hopefully reducing the use of traditional chemotherapy in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Females ≥ 18 years old at the time of the ICF signature
* histologically confirmed locally advanced breast carcinoma, defined as either large T2 (>3cm in diameter) or T3-T4, and/or N2-3 primary breast cancer
* ER-positive (defined by ER-pos. in ≥ 50% of cancer cells) and HER-2 negative, luminal A/B breast cancer
* postmenopausal status (natural status or induced by treatment with the LHRH-analogue goserelin 3.6mg implant s.c. given every 4 weeks); definition of natural post-menopausal status: age above 55 years or age above 50 years and at least 2 years of amenorrhea in addition to LH-, FSH-, and plasma estradiol levels in the post-menopausal range.
* Patient has adequate bone marrow and organ function as defined by the following laboratory values (as assessed by central laboratory eligibility): Absolute neutrophil count ≥ 1.0x109/L; platelets ≥ 100 x 109/L; Hemoglobin ≥ 9.0g/dL; INR≤1.5 (unless the patient is receiving anticoagulants and the INR is within the therapeutic range of intended use for that anticoagulant within 7 days prior to the first dose of study drug); Estimated glomerular filtration rate (eGFR) ≥ 30mL/min/1.73m2 according to the Modification of Diet in Renal Disease (MDRD) formula; total bilirubin < ULN except for patients with Gilbert's syndrome who may only be included if the total bilirubin is ≤ 3.0 x ULN or direct bilirubin ≤ 1.5 x ULN; aspartate transaminase (AST) < 2.5 x ULN; Alanine transaminase (ALT) < 2.5 x ULN; patient must have the following laboratory values within normal limits or corrected to within normal limits with supplements before the first dose of study medication: potassium, magnesium, total calcium (corrected for serum albumin).
* Standard 12-lead ECG values defined as the mean of the triplicate ECGs [QTcF interval at screening < 450 msec (QT interval using Fridericia's correction), mean resting heart rate 50-90 bpm (determined from the ECG)]
* Performance status: Eastern Cooperative Oncology Group (ECOG) score 0-1
* Ability and willingness to comply with study visits, treatment, testing and to comply with the protocol.

Exclusion Criteria:

* Any prior treatment for primary invasive breast cancer
* Patient with a known hypersensitivity to any of the excipients of ribociclib or letrozole
* Patient with known hypersensitivity to peanuts or soya-products
* Any evidence of distant metastasis
* Triple-negative breast cancer
* HER-2 positive disease, suitable for neoadjuvant therapy with trastuzumab, pertuzumab and taxanes, etc.
* Other conditions rendering patients in need of other treatment options with immediate effect like chemotherapy
* Concomitant medications that are known strong inducers of CYP3A4/5
* Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality, including any of the following: History of documented myocardial infarction (MI), angina pectoris, symptomatic pericarditis, or coronary artery bypass graft (CABG) within 6 months prior to study entry; documented cardiomyopathy; Left Ventricular Ejection Fraction (LVEF) < 50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO); Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following: Risk factors for Torsades de Pointe (TdP) including uncorrected hypocalcemia, hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia, Concomitant medication(s) with a known risk to prolong the QT interval and/or known to cause Torsades de Pointe that cannot be discontinued or replaced by safe alternative medication (e.g., within 5 half-lives or 7 days prior to starting study drug) or Inability to determine the QTcF interval; Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g., bifascicular block, Mobitz type II and third degree AV block); Systolic Blood Pressure (SBP) >160 or <90 mmHg
* Patient is currently receiving or has received systemic corticosteroids ≤ 2 weeks prior to starting study drug, or who have not fully recovered from side effects of such treatment. Note: The following uses of corticosteroids are permitted: a short duration (<5 days) of systemic corticosteroids; any duration of topical applications (e.g. for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intraarticular).
* Pregnant or breast-feeding (lactating) women or women who plan to become pregnant or breast-feed during the trial
* Women of child-bearing potential defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during the study treatment and for 21 days after stopping the treatment. Highly effective contraception methods include: Total abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception; Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or tubal ligation at least 6 weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment; Male partner sterilization (at least 6 months prior to screening). For female patients on the study, the vasectomized male partner should be the sole partner for that patient and the success of the vasectomy must be medically confirmed as per local practice; Placement of an intrauterine device (IUD); Note: Use of oral (estrogen and progesterone), transdermal, injected, implanted, hormone containing intrauterine systems (IUS) or any other hormonal methods of contraception is not allowed in this study
* Autoimmune disorders or significant allergies (i.e. rheumatoid arthritis, asthma, psoriasis, etc.)
* Known HIV infection, Hepatitis B or C infection (testing not mandatory)
* History of autoimmune celiac, inflammatory bowel disease, or other chronic GI disease
* Recent use (within past month) of more than 3 days of antibiotics use
* Current use of probiotic supplements
* Taking proton pump inhibitors, steroids, other non-steroidal antiinflammatory drugs such as ibuprofen or acetyl salicylic acid
* Past bariatric surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
To study the change in levels of direct and indirect immunologic biomarkers of targeted cancer therapy with letrozole and ribociclib given in combination for patients with locally-advanced, ER-positive, HER-2 negative, luminal A7B breast cancer | Baseline, Day 21 and at time of surgery (Day 180)
  In order to accurately profile changes in the composition of the tumor over time and identify potentially-related biomarkers of response within the tumor, single cell RNA panels will be performed at three points during the treatment period. Samples of tumor tissue will be obtained, and the cells dissociated at the single cell level. These dissociated cells will then be subjected to RNA profiling via scRNA-seq. Genes expressed at a rate higher than the threshhold (generally 50 reads per kb per million reads) will be examined using t-Distributed Stochastic Neighbor Embedding, (tSNE) clustering, generally shown as a scatterplot, to allow the characterisation of phenotypes (clones). Using this technique, it will be evident which tumour phenotypes are eradicated by the treatment combination and which are not. This examination will also help to monitor patient response.

SECONDARY OUTCOMES:
Measurement of changes in the tumor through DNA profiling throughout the treatment cycle with letrozole and ribociclib | Baseline, Day 21 and at time of surgery (Day 180)
  In order to examine the potential genetic changes within the tumor during treatment, samples of tumor tissue will be taken and examined using standard DNA profiling. Baseline samples will be compared to those at day 21 and at the time of surgery (6 months). This outcome will allow identification of overall tumour composition and changes to over the course of the therapy.
Confirmation of the breast cancer subtype | Baseline
  To determine the subtypes of the tumor, a PROSIGNA-test will be undertaken on all samples to confirm their subtype.
Changes in neoantigens and single T-cell receptor function after treatment with letrozole and ribociclib | Baseline, Day 21 and at time of surgery (Day 180)
  In order to examine the effects of letrozole and ribociclib on the presence of immune cells within the tumor throughout treatment, samples of tumor tissue will be extracted and cells will be dissociated at the single-cell level using enzymatic and mechanical means. Measurement of tumor neoantigens and testing of the ability of the T-cell receptors to recognise these neoantigens will assist in the understanding of the "rules" and molecular events underlying immune-mediated tumor destruction. Further, responders and non-responders will be compared to identify whether they belong to a new yet undiscovered subtype.
Determination of the histopathological sub-type and status of the tumour | Baseline, Day 21 and at time of surgery (Day 180)
  To ensure the correct patients are identified for participation in this study, and to record overall baseline information, samples of tumor tissue will be examined via standard histopathological investigations including subtyping, grading, ER-status, PGR-status, HER-2 status and level of Ki67-expression will be undertaken by a qualified pathologist. After the baseline, examination will confirm that biopsies consist of tumor tissue.
Determination of the early and late mechanisms of adaptation and/or resistance to letrozole in combination with ribociclib | Baseline and at time of surgery (Day 180)
  Using single-cell RNA-seq (scRNA-seq), thousands of individual cells will be profiled to build a cellular atlas of whole tumor biomarkers for targeted cancer treatments. scRNA-seq allows the characterisation of phenotypes (clones) to assist in determination of the phenotypes eradicated by the treatment, and to find biomarkers of response. Further knowledge of the phenotypes of the cells most affected by the therapy may assist in the identification of further drugs targeting any cells that remain or thrive.
Change in PEPI status from baseline in response to targeted neoadjuvant therapy with letrozole and ribociclib | Baseline, Day 21, Day 90, Day 180
  Preoperative endocrine prognostic index (PEPI) status will be evaluated across the treatment period using the procedure outlined in Ellis et al, 2008.
Change in Ki67 from baseline in response to targeted neoadjuvant therapy with letrozole and ribociclib | Baseline, Day 21, Day 90, Day 180
  Levels of Ki67 will be evaluated across the study period using the XXXXX protocol. Complete Cell Cycle Arrest (CCCA) will be recorded as a Ki67 of less than 2.7%.
Change in PROSIGNA Risk of Recurrence (ROR) score from baseline in response to targeted neoadjuvant therapy with letrozole and ribociclib | Baseline, Day 21, Day 90, Day 180
Changes in the composition of the gut microbiota | Baseline, 21 and 90, at time of surgery (Day 180), and annually in years 1-5 (extension if patient relapses)
  A DNA-based approach to determination of fecal microbial composition will be performed. Stool samples will be collected at baseline, and during follow ups at day 21, day 90 and at time of surgery (day 180), and thereafter annually in years 1-5 (further if patient relapses). DNA purification from fecal samples will be performed using PSP Spin Stool DNA Plus Kit (Stratec Molecular GMBH). Next generation amplicon sequencing targeting the V4 region of the 16S rRNA gene (DNA) will be applied to detect the members of the fecal microbiota.
Identification of anti-tumor effects via changes in levels of circulating serum cytokines in liquid biopsies | Baseline, 21 and 90, and at time of surgery (Day 180).
  Serum cytokines will be measured using 54-plex cytokine panel, and analyzed with Luminex xMAP 200. The assay includes a series of known concentrations giving standard curves. Samples will be analyzed in duplicate.
Identification of anti-tumor effects via changes in levels of circulating serum metabolites in liquid biopsies | Baseline, 21 and 90, and at time of surgery (Day 180).
  Circulating metabolites will be identified using high resolution magic angle spinning mass spectrometry as described in Bathen et al (2013).
Identification of anti-tumor effects via circulating free tumor DNA (cftDNA) in liquid biopsies | Baseline, 21 and 90, and at time of surgery (Day 180).
  Circulating free tumor DNA will be collected and identified using standard DNA extraction and analysis techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Geisler, MD, PhD, Principal Investigator — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Lørenskog, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No
Norwegian data protection laws are very strict, and free access to patient data is not possible. Authorised Norwegian researchers who wish to gain access to the data may apply individually to the study PI.

REFERENCES:
- [Background] Semiglazov VF, Semiglazov VV, Dashyan GA, Ziltsova EK, Ivanov VG, Bozhok AA, Melnikova OA, Paltuev RM, Kletzel A, Berstein LM. Phase 2 randomized trial of primary endocrine therapy versus chemotherapy in postmenopausal patients with estrogen receptor-positive breast cancer. Cancer. 2007 Jul 15;110(2):244-54. doi: 10.1002/cncr.22789. PMID 17538978
- [Background] Smith IE, Dowsett M, Ebbs SR, Dixon JM, Skene A, Blohmer JU, Ashley SE, Francis S, Boeddinghaus I, Walsh G; IMPACT Trialists Group. Neoadjuvant treatment of postmenopausal breast cancer with anastrozole, tamoxifen, or both in combination: the Immediate Preoperative Anastrozole, Tamoxifen, or Combined with Tamoxifen (IMPACT) multicenter double-blind randomized trial. J Clin Oncol. 2005 Aug 1;23(22):5108-16. doi: 10.1200/JCO.2005.04.005. Epub 2005 Jul 5. PMID 15998903
- [Background] Geisler J, Detre S, Berntsen H, Ottestad L, Lindtjorn B, Dowsett M, Einstein Lonning P. Influence of neoadjuvant anastrozole (Arimidex) on intratumoral estrogen levels and proliferation markers in patients with locally advanced breast cancer. Clin Cancer Res. 2001 May;7(5):1230-6. PMID 11350888
- [Background] Geisler J, Haynes B, Anker G, Dowsett M, Lonning PE. Influence of letrozole and anastrozole on total body aromatization and plasma estrogen levels in postmenopausal breast cancer patients evaluated in a randomized, cross-over study. J Clin Oncol. 2002 Feb 1;20(3):751-7. doi: 10.1200/JCO.2002.20.3.751. PMID 11821457
- [Background] Geisler J, Helle H, Ekse D, Duong NK, Evans DB, Nordbo Y, Aas T, Lonning PE. Letrozole is superior to anastrozole in suppressing breast cancer tissue and plasma estrogen levels. Clin Cancer Res. 2008 Oct 1;14(19):6330-5. doi: 10.1158/1078-0432.CCR-07-5221. PMID 18829517
- [Background] Geisler J, King N, Anker G, Ornati G, Di Salle E, Lonning PE, Dowsett M. In vivo inhibition of aromatization by exemestane, a novel irreversible aromatase inhibitor, in postmenopausal breast cancer patients. Clin Cancer Res. 1998 Sep;4(9):2089-93. PMID 9748124
- [Background] Geisler J, King N, Dowsett M, Ottestad L, Lundgren S, Walton P, Kormeset PO, Lonning PE. Influence of anastrozole (Arimidex), a selective, non-steroidal aromatase inhibitor, on in vivo aromatisation and plasma oestrogen levels in postmenopausal women with breast cancer. Br J Cancer. 1996 Oct;74(8):1286-91. doi: 10.1038/bjc.1996.531. PMID 8883419
- [Background] Gnant M, Steger GG, Bartsch R. CDK4/6 inhibitors in luminal breast cancer. Lancet Oncol. 2015 Jan;16(1):2-3. doi: 10.1016/S1470-2045(14)71188-X. Epub 2014 Dec 16. No abstract available. PMID 25524801
- [Background] Lim JS, Turner NC, Yap TA. CDK4/6 Inhibitors: Promising Opportunities beyond Breast Cancer. Cancer Discov. 2016 Jul;6(7):697-9. doi: 10.1158/2159-8290.CD-16-0563. PMID 27371575
- [Background] Hortobagyi GN, Stemmer SM, Burris HA, Yap YS, Sonke GS, Paluch-Shimon S, Campone M, Petrakova K, Blackwell KL, Winer EP, Janni W, Verma S, Conte P, Arteaga CL, Cameron DA, Mondal S, Su F, Miller M, Elmeliegy M, Germa C, O'Shaughnessy J. Updated results from MONALEESA-2, a phase III trial of first-line ribociclib plus letrozole versus placebo plus letrozole in hormone receptor-positive, HER2-negative advanced breast cancer. Ann Oncol. 2018 Jul 1;29(7):1541-1547. doi: 10.1093/annonc/mdy155. PMID 29718092
- [Background] Hortobagyi GN, Stemmer SM, Burris HA, Yap YS, Sonke GS, Paluch-Shimon S, Campone M, Petrakova K, Blackwell KL, Winer EP, Janni W, Verma S, Conte P, Arteaga CL, Cameron DA, Mondal S, Su F, Miller M, Elmeliegy M, Germa C, O'Shaughnessy J. Updated results from MONALEESA-2, a phase III trial of first-line ribociclib plus letrozole versus placebo plus letrozole in hormone receptor-positive, HER2-negative advanced breast cancer. Ann Oncol. 2019 Nov 1;30(11):1842. doi: 10.1093/annonc/mdz215. No abstract available. PMID 31407010
- [Background] Finn RS, Martin M, Rugo HS, Jones S, Im SA, Gelmon K, Harbeck N, Lipatov ON, Walshe JM, Moulder S, Gauthier E, Lu DR, Randolph S, Dieras V, Slamon DJ. Palbociclib and Letrozole in Advanced Breast Cancer. N Engl J Med. 2016 Nov 17;375(20):1925-1936. doi: 10.1056/NEJMoa1607303. PMID 27959613
- [Background] Slamon DJ, Neven P, Chia S, Fasching PA, De Laurentiis M, Im SA, Petrakova K, Bianchi GV, Esteva FJ, Martin M, Nusch A, Sonke GS, De la Cruz-Merino L, Beck JT, Pivot X, Vidam G, Wang Y, Rodriguez Lorenc K, Miller M, Taran T, Jerusalem G. Phase III Randomized Study of Ribociclib and Fulvestrant in Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Advanced Breast Cancer: MONALEESA-3. J Clin Oncol. 2018 Aug 20;36(24):2465-2472. doi: 10.1200/JCO.2018.78.9909. Epub 2018 Jun 3. PMID 29860922
- [Background] Turner NC, Ro J, Andre F, Loi S, Verma S, Iwata H, Harbeck N, Loibl S, Huang Bartlett C, Zhang K, Giorgetti C, Randolph S, Koehler M, Cristofanilli M; PALOMA3 Study Group. Palbociclib in Hormone-Receptor-Positive Advanced Breast Cancer. N Engl J Med. 2015 Jul 16;373(3):209-19. doi: 10.1056/NEJMoa1505270. Epub 2015 Jun 1. PMID 26030518
- [Background] Cristofanilli M, Turner NC, Bondarenko I, Ro J, Im SA, Masuda N, Colleoni M, DeMichele A, Loi S, Verma S, Iwata H, Harbeck N, Zhang K, Theall KP, Jiang Y, Bartlett CH, Koehler M, Slamon D. Fulvestrant plus palbociclib versus fulvestrant plus placebo for treatment of hormone-receptor-positive, HER2-negative metastatic breast cancer that progressed on previous endocrine therapy (PALOMA-3): final analysis of the multicentre, double-blind, phase 3 randomised controlled trial. Lancet Oncol. 2016 Apr;17(4):425-439. doi: 10.1016/S1470-2045(15)00613-0. Epub 2016 Mar 3. PMID 26947331
- [Background] Turner NC, Slamon DJ, Ro J, Bondarenko I, Im SA, Masuda N, Colleoni M, DeMichele A, Loi S, Verma S, Iwata H, Harbeck N, Loibl S, Andre F, Puyana Theall K, Huang X, Giorgetti C, Huang Bartlett C, Cristofanilli M. Overall Survival with Palbociclib and Fulvestrant in Advanced Breast Cancer. N Engl J Med. 2018 Nov 15;379(20):1926-1936. doi: 10.1056/NEJMoa1810527. Epub 2018 Oct 20. PMID 30345905
- [Background] McCaw ZR, Vassy JL, Wei LJ. Palbociclib and Fulvestrant in Breast Cancer. N Engl J Med. 2019 Feb 21;380(8):796. doi: 10.1056/NEJMc1816595. No abstract available. PMID 30789681
- [Background] Prat A, Saura C, Pascual T, Hernando C, Munoz M, Pare L, Gonzalez Farre B, Fernandez PL, Galvan P, Chic N, Gonzalez Farre X, Oliveira M, Gil-Gil M, Arumi M, Ferrer N, Montano A, Izarzugaza Y, Llombart-Cussac A, Bratos R, Gonzalez Santiago S, Martinez E, Hoyos S, Rojas B, Virizuela JA, Ortega V, Lopez R, Celiz P, Ciruelos E, Villagrasa P, Gavila J. Ribociclib plus letrozole versus chemotherapy for postmenopausal women with hormone receptor-positive, HER2-negative, luminal B breast cancer (CORALLEEN): an open-label, multicentre, randomised, phase 2 trial. Lancet Oncol. 2020 Jan;21(1):33-43. doi: 10.1016/S1470-2045(19)30786-7. Epub 2019 Dec 11. PMID 31838010
- [Background] Slamon DJ, Neven P, Chia S, Fasching PA, De Laurentiis M, Im SA, Petrakova K, Bianchi GV, Esteva FJ, Martin M, Nusch A, Sonke GS, De la Cruz-Merino L, Beck JT, Pivot X, Sondhi M, Wang Y, Chakravartty A, Rodriguez-Lorenc K, Taran T, Jerusalem G. Overall Survival with Ribociclib plus Fulvestrant in Advanced Breast Cancer. N Engl J Med. 2020 Feb 6;382(6):514-524. doi: 10.1056/NEJMoa1911149. Epub 2019 Dec 11. PMID 31826360
- [Background] Rocca A, Melegari E, Palleschi M. Ribociclib and Endocrine Therapy in Breast Cancer. N Engl J Med. 2019 Oct 17;381(16):1592. doi: 10.1056/NEJMc1911188. No abstract available. PMID 31618549
- [Background] Im SA, Lu YS, Bardia A, Harbeck N, Colleoni M, Franke F, Chow L, Sohn J, Lee KS, Campos-Gomez S, Villanueva-Vazquez R, Jung KH, Chakravartty A, Hughes G, Gounaris I, Rodriguez-Lorenc K, Taran T, Hurvitz S, Tripathy D. Overall Survival with Ribociclib plus Endocrine Therapy in Breast Cancer. N Engl J Med. 2019 Jul 25;381(4):307-316. doi: 10.1056/NEJMoa1903765. Epub 2019 Jun 4. PMID 31166679
- [Background] Johnston S, Puhalla S, Wheatley D, Ring A, Barry P, Holcombe C, Boileau JF, Provencher L, Robidoux A, Rimawi M, McIntosh SA, Shalaby I, Stein RC, Thirlwell M, Dolling D, Morden J, Snowdon C, Perry S, Cornman C, Batten LM, Jeffs LK, Dodson A, Martins V, Modi A, Osborne CK, Pogue-Geile KL, Cheang MCU, Wolmark N, Julian TB, Fisher K, MacKenzie M, Wilcox M, Huang Bartlett C, Koehler M, Dowsett M, Bliss JM, Jacobs SA. Randomized Phase II Study Evaluating Palbociclib in Addition to Letrozole as Neoadjuvant Therapy in Estrogen Receptor-Positive Early Breast Cancer: PALLET Trial. J Clin Oncol. 2019 Jan 20;37(3):178-189. doi: 10.1200/JCO.18.01624. Epub 2018 Dec 6. PMID 30523750
- [Background] Gianni L, Bisagni G, Colleoni M, Del Mastro L, Zamagni C, Mansutti M, Zambetti M, Frassoldati A, De Fato R, Valagussa P, Viale G. Neoadjuvant treatment with trastuzumab and pertuzumab plus palbociclib and fulvestrant in HER2-positive, ER-positive breast cancer (NA-PHER2): an exploratory, open-label, phase 2 study. Lancet Oncol. 2018 Feb;19(2):249-256. doi: 10.1016/S1470-2045(18)30001-9. Epub 2018 Jan 8. PMID 29326029
- [Background] Cottu P, D'Hondt V, Dureau S, Lerebours F, Desmoulins I, Heudel PE, Duhoux FP, Levy C, Mouret-Reynier MA, Dalenc F, Frenel JS, Jouannaud C, Venat-Bouvet L, Nguyen S, Ferrero JM, Canon JL, Grenier J, Callens C, Gentien D, Lemonnier J, Vincent-Salomon A, Delaloge S. Letrozole and palbociclib versus chemotherapy as neoadjuvant therapy of high-risk luminal breast cancer. Ann Oncol. 2018 Dec 1;29(12):2334-2340. doi: 10.1093/annonc/mdy448. PMID 30307466
- [Background] Chow LWC, Morita S, Chow CYC, Ng WK, Toi M. Neoadjuvant palbociclib on ER+ breast cancer (N007): clinical response and EndoPredict's value. Endocr Relat Cancer. 2018 Feb;25(2):123-130. doi: 10.1530/ERC-17-0396. Epub 2017 Nov 20. PMID 29158285
- [Background] Ma CX, Gao F, Luo J, Northfelt DW, Goetz M, Forero A, Hoog J, Naughton M, Ademuyiwa F, Suresh R, Anderson KS, Margenthaler J, Aft R, Hobday T, Moynihan T, Gillanders W, Cyr A, Eberlein TJ, Hieken T, Krontiras H, Guo Z, Lee MV, Spies NC, Skidmore ZL, Griffith OL, Griffith M, Thomas S, Bumb C, Vij K, Bartlett CH, Koehler M, Al-Kateb H, Sanati S, Ellis MJ. NeoPalAna: Neoadjuvant Palbociclib, a Cyclin-Dependent Kinase 4/6 Inhibitor, and Anastrozole for Clinical Stage 2 or 3 Estrogen Receptor-Positive Breast Cancer. Clin Cancer Res. 2017 Aug 1;23(15):4055-4065. doi: 10.1158/1078-0432.CCR-16-3206. Epub 2017 Mar 7. PMID 28270497
- [Background] Buyukkaramikli NC, de Groot S, Riemsma R, Fayter D, Armstrong N, Portegijs P, Duffy S, Kleijnen J, Al MJ. Ribociclib with an Aromatase Inhibitor for Previously Untreated, HR-Positive, HER2-Negative, Locally Advanced or Metastatic Breast Cancer: An Evidence Review Group Perspective of a NICE Single Technology Appraisal. Pharmacoeconomics. 2019 Feb;37(2):141-153. doi: 10.1007/s40273-018-0708-4. PMID 30194622
- [Background] Tekpli X, Lien T, Rossevold AH, Nebdal D, Borgen E, Ohnstad HO, Kyte JA, Vallon-Christersson J, Fongaard M, Due EU, Svartdal LG, Sveli MAT, Garred O; OSBREAC; Frigessi A, Sahlberg KK, Sorlie T, Russnes HG, Naume B, Kristensen VN. An independent poor-prognosis subtype of breast cancer defined by a distinct tumor immune microenvironment. Nat Commun. 2019 Dec 3;10(1):5499. doi: 10.1038/s41467-019-13329-5. PMID 31796750
- [Background] Jabeen S, Zucknick M, Nome M, Dannenfelser R, Fleischer T, Kumar S, Luders T, von der Lippe Gythfeldt H, Troyanskaya O, Kyte JA, Borresen-Dale AL, Naume B, Tekpli X, Engebraaten O, Kristensen V. Serum cytokine levels in breast cancer patients during neoadjuvant treatment with bevacizumab. Oncoimmunology. 2018 Aug 6;7(11):e1457598. doi: 10.1080/2162402X.2018.1457598. eCollection 2018. PMID 30377556
- [Background] Vetizou M, Pitt JM, Daillere R, Lepage P, Waldschmitt N, Flament C, Rusakiewicz S, Routy B, Roberti MP, Duong CP, Poirier-Colame V, Roux A, Becharef S, Formenti S, Golden E, Cording S, Eberl G, Schlitzer A, Ginhoux F, Mani S, Yamazaki T, Jacquelot N, Enot DP, Berard M, Nigou J, Opolon P, Eggermont A, Woerther PL, Chachaty E, Chaput N, Robert C, Mateus C, Kroemer G, Raoult D, Boneca IG, Carbonnel F, Chamaillard M, Zitvogel L. Anticancer immunotherapy by CTLA-4 blockade relies on the gut microbiota. Science. 2015 Nov 27;350(6264):1079-84. doi: 10.1126/science.aad1329. Epub 2015 Nov 5. PMID 26541610
- [Background] Elkrief A, Derosa L, Zitvogel L, Kroemer G, Routy B. The intimate relationship between gut microbiota and cancer immunotherapy. Gut Microbes. 2019;10(3):424-428. doi: 10.1080/19490976.2018.1527167. Epub 2018 Oct 19. PMID 30339501
- [Background] Routy B, Gopalakrishnan V, Daillere R, Zitvogel L, Wargo JA, Kroemer G. The gut microbiota influences anticancer immunosurveillance and general health. Nat Rev Clin Oncol. 2018 Jun;15(6):382-396. doi: 10.1038/s41571-018-0006-2. PMID 29636538
- [Background] Kroemer G, Zitvogel L. Cancer immunotherapy in 2017: The breakthrough of the microbiota. Nat Rev Immunol. 2018 Jan 30;18(2):87-88. doi: 10.1038/nri.2018.4. No abstract available. PMID 29379189
- [Background] Chew CS. Parietal cell protein kinases. Selective activation of type I cAMP-dependent protein kinase by histamine. J Biol Chem. 1985 Jun 25;260(12):7540-50. PMID 2987257
- [Background] Zitvogel L, Galluzzi L, Viaud S, Vetizou M, Daillere R, Merad M, Kroemer G. Cancer and the gut microbiota: an unexpected link. Sci Transl Med. 2015 Jan 21;7(271):271ps1. doi: 10.1126/scitranslmed.3010473. PMID 25609166
- [Background] Viaud S, Saccheri F, Mignot G, Yamazaki T, Daillere R, Hannani D, Enot DP, Pfirschke C, Engblom C, Pittet MJ, Schlitzer A, Ginhoux F, Apetoh L, Chachaty E, Woerther PL, Eberl G, Berard M, Ecobichon C, Clermont D, Bizet C, Gaboriau-Routhiau V, Cerf-Bensussan N, Opolon P, Yessaad N, Vivier E, Ryffel B, Elson CO, Dore J, Kroemer G, Lepage P, Boneca IG, Ghiringhelli F, Zitvogel L. The intestinal microbiota modulates the anticancer immune effects of cyclophosphamide. Science. 2013 Nov 22;342(6161):971-6. doi: 10.1126/science.1240537. PMID 24264990
- [Background] Gopalakrishnan V, Spencer CN, Nezi L, Reuben A, Andrews MC, Karpinets TV, Prieto PA, Vicente D, Hoffman K, Wei SC, Cogdill AP, Zhao L, Hudgens CW, Hutchinson DS, Manzo T, Petaccia de Macedo M, Cotechini T, Kumar T, Chen WS, Reddy SM, Szczepaniak Sloane R, Galloway-Pena J, Jiang H, Chen PL, Shpall EJ, Rezvani K, Alousi AM, Chemaly RF, Shelburne S, Vence LM, Okhuysen PC, Jensen VB, Swennes AG, McAllister F, Marcelo Riquelme Sanchez E, Zhang Y, Le Chatelier E, Zitvogel L, Pons N, Austin-Breneman JL, Haydu LE, Burton EM, Gardner JM, Sirmans E, Hu J, Lazar AJ, Tsujikawa T, Diab A, Tawbi H, Glitza IC, Hwu WJ, Patel SP, Woodman SE, Amaria RN, Davies MA, Gershenwald JE, Hwu P, Lee JE, Zhang J, Coussens LM, Cooper ZA, Futreal PA, Daniel CR, Ajami NJ, Petrosino JF, Tetzlaff MT, Sharma P, Allison JP, Jenq RR, Wargo JA. Gut microbiome modulates response to anti-PD-1 immunotherapy in melanoma patients. Science. 2018 Jan 5;359(6371):97-103. doi: 10.1126/science.aan4236. Epub 2017 Nov 2. PMID 29097493
- [Background] Kala M, Chrobok J, Dvorak P. A surprising finding by a surgery for lumbar intervertebral disk herniation--Ewing's sarcoma. Acta Univ Palacki Olomuc Fac Med. 1987;117:185-9. No abstract available. PMID 2963494
- [Background] Routy B, Le Chatelier E, Derosa L, Duong CPM, Alou MT, Daillere R, Fluckiger A, Messaoudene M, Rauber C, Roberti MP, Fidelle M, Flament C, Poirier-Colame V, Opolon P, Klein C, Iribarren K, Mondragon L, Jacquelot N, Qu B, Ferrere G, Clemenson C, Mezquita L, Masip JR, Naltet C, Brosseau S, Kaderbhai C, Richard C, Rizvi H, Levenez F, Galleron N, Quinquis B, Pons N, Ryffel B, Minard-Colin V, Gonin P, Soria JC, Deutsch E, Loriot Y, Ghiringhelli F, Zalcman G, Goldwasser F, Escudier B, Hellmann MD, Eggermont A, Raoult D, Albiges L, Kroemer G, Zitvogel L. Gut microbiome influences efficacy of PD-1-based immunotherapy against epithelial tumors. Science. 2018 Jan 5;359(6371):91-97. doi: 10.1126/science.aan3706. Epub 2017 Nov 2. PMID 29097494
- [Background] Ebert PJR, Cheung J, Yang Y, McNamara E, Hong R, Moskalenko M, Gould SE, Maecker H, Irving BA, Kim JM, Belvin M, Mellman I. MAP Kinase Inhibition Promotes T Cell and Anti-tumor Activity in Combination with PD-L1 Checkpoint Blockade. Immunity. 2016 Mar 15;44(3):609-621. doi: 10.1016/j.immuni.2016.01.024. Epub 2016 Mar 2. PMID 26944201
- [Background] Deng J, Wang ES, Jenkins RW, Li S, Dries R, Yates K, Chhabra S, Huang W, Liu H, Aref AR, Ivanova E, Paweletz CP, Bowden M, Zhou CW, Herter-Sprie GS, Sorrentino JA, Bisi JE, Lizotte PH, Merlino AA, Quinn MM, Bufe LE, Yang A, Zhang Y, Zhang H, Gao P, Chen T, Cavanaugh ME, Rode AJ, Haines E, Roberts PJ, Strum JC, Richards WG, Lorch JH, Parangi S, Gunda V, Boland GM, Bueno R, Palakurthi S, Freeman GJ, Ritz J, Haining WN, Sharpless NE, Arthanari H, Shapiro GI, Barbie DA, Gray NS, Wong KK. CDK4/6 Inhibition Augments Antitumor Immunity by Enhancing T-cell Activation. Cancer Discov. 2018 Feb;8(2):216-233. doi: 10.1158/2159-8290.CD-17-0915. Epub 2017 Nov 3. PMID 29101163
- [Background] Goel S, DeCristo MJ, Watt AC, BrinJones H, Sceneay J, Li BB, Khan N, Ubellacker JM, Xie S, Metzger-Filho O, Hoog J, Ellis MJ, Ma CX, Ramm S, Krop IE, Winer EP, Roberts TM, Kim HJ, McAllister SS, Zhao JJ. CDK4/6 inhibition triggers anti-tumour immunity. Nature. 2017 Aug 24;548(7668):471-475. doi: 10.1038/nature23465. Epub 2017 Aug 16. PMID 28813415
- [Background] Zhang J, Bu X, Wang H, Zhu Y, Geng Y, Nihira NT, Tan Y, Ci Y, Wu F, Dai X, Guo J, Huang YH, Fan C, Ren S, Sun Y, Freeman GJ, Sicinski P, Wei W. Cyclin D-CDK4 kinase destabilizes PD-L1 via cullin 3-SPOP to control cancer immune surveillance. Nature. 2018 Jan 4;553(7686):91-95. doi: 10.1038/nature25015. Epub 2017 Nov 16. PMID 29160310
- [Background] Petroni G, Formenti SC, Chen-Kiang S, Galluzzi L. Immunomodulation by anticancer cell cycle inhibitors. Nat Rev Immunol. 2020 Nov;20(11):669-679. doi: 10.1038/s41577-020-0300-y. Epub 2020 Apr 28. PMID 32346095
- [Background] Goel S, Tolaney SM. CDK4/6 inhibitors in breast cancer: a role in triple-negative disease? Lancet Oncol. 2019 Nov;20(11):1479-1481. doi: 10.1016/S1470-2045(19)30627-8. Epub 2019 Sep 28. No abstract available. PMID 31575504
- [Background] Wang L, Ellsworth KA, Moon I, Pelleymounter LL, Eckloff BW, Martin YN, Fridley BL, Jenkins GD, Batzler A, Suman VJ, Ravi S, Dixon JM, Miller WR, Wieben ED, Buzdar A, Weinshilboum RM, Ingle JN. Functional genetic polymorphisms in the aromatase gene CYP19 vary the response of breast cancer patients to neoadjuvant therapy with aromatase inhibitors. Cancer Res. 2010 Jan 1;70(1):319-28. doi: 10.1158/0008-5472.CAN-09-3224. PMID 20048079
- [Background] Geisler J, Smith I, Miller W. Presurgical (neoadjuvant) endocrine therapy is a useful model to predict response and outcome to endocrine treatment in breast cancer patients. J Steroid Biochem Mol Biol. 2012 Sep;131(3-5):93-100. doi: 10.1016/j.jsbmb.2011.12.006. Epub 2011 Dec 22. PMID 22207086
- [Background] Bathen TF, Geurts B, Sitter B, Fjosne HE, Lundgren S, Buydens LM, Gribbestad IS, Postma G, Giskeodegard GF. Feasibility of MR metabolomics for immediate analysis of resection margins during breast cancer surgery. PLoS One. 2013 Apr 17;8(4):e61578. doi: 10.1371/journal.pone.0061578. Print 2013. PMID 23613877
- [Background] Ellis MJ, Tao Y, Luo J, A'Hern R, Evans DB, Bhatnagar AS, Chaudri Ross HA, von Kameke A, Miller WR, Smith I, Eiermann W, Dowsett M. Outcome prediction for estrogen receptor-positive breast cancer based on postneoadjuvant endocrine therapy tumor characteristics. J Natl Cancer Inst. 2008 Oct 1;100(19):1380-8. doi: 10.1093/jnci/djn309. Epub 2008 Sep 23. PMID 18812550
- [Derived] Fjermeros K, Ghannoum S, Geisler SB, Bhargava S, Tahiri A, Klajic J, Luders T, Fongard M, Nawaz MS, Bosnjak-Olsen T, Buvarp UE, Rosenskiold AKJ, Nguyen NT, Sletbak TT, Seyedzadeh M, Selsas K, Porojnicu AC, Skjerven HK, Hovda T, Sahlberg KK, Torland LA, Lyngra M, Hammarstrom CL, Honigsperger EB, Noone JC, Mathiassen S, Hurtado A, Goel S, Koff A, Tekpli X, Kristensen VN, Geisler J. The NEOLETRIB trial: neoadjuvant treatment with Letrozole and Ribociclib in ER-positive, HER2-negative breast cancer. Future Oncol. 2024;20(32):2457-2466. doi: 10.1080/14796694.2024.2377531. Epub 2024 Jul 29. PMID 39073142

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT05163106/Prot_SAP_000.pdf